CLINICAL TRIAL: NCT02189538
Title: Effect of Omega-3 PUFA From Fish in Major Burn Patients. EFECTO DE ÁCIDOS GRASOS POLIINSATURADOS OMEGA 3 DERIVADOS DE ACEITE DE PESCADO, EN QUEMADOS GRAVES
Brief Title: Effect of n-3 PUFA From Fish in Enteral Nutrition of Major Burn Patients
Acronym: OmegaBurn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Nacional de Quemados, Uruguay (Other)
Responsible Party: Principal Investigator, Serrana Tihista, dietitian, Centro Nacional de Quemados, Uruguay
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Universidad de la República
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-02

CONDITIONS: Burn Injury
Keywords: Infections, Enteral nutrition, SIRS, critically ill
MeSH Terms: conditions — Burns; Infections; Critical Illness | interventions — CD36 Antigens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ω-3 PUFA (Experimental): Modular low fat diet (18%) including 9% as ω-3 PUFA
  Interventions: Dietary Supplement: ω-3 PUFA
- Low fat enteral diet (Active Comparator): Modular low fat (18%)
  Interventions: Dietary Supplement: Low fat enteral diet

INTERVENTIONS:
Dietary Supplement: ω-3 PUFA — The patients are fed as long as the clinically required with the randomly attributed enteral solution.
  Other Names: modular preparation: 9% ω-3 of the total 18% fat
  Arms: ω-3 PUFA
Dietary Supplement: Low fat enteral diet — The patients are fed as long as the clinically required with the randomly attributed enteral solution
  Other Names: modular diet
  Arms: Low fat enteral diet

SUMMARY:
Studies have shown that burn patients may benefit from low fat diets, but there is still no strong data regarding the impact of fatty acid composition used for feeding. The trial test the hypothesis that the inclusion of omega-3 PUFA in a low fat diet may improve outcome. Prospective randomised controlled trial in adult patients admitted for burns > 15% body surface area (BSA), and inhalation injury requiring mechanical ventilation and enteral nutrition. On admission randomization to receive a low-fat (18% energy as fat) modular enteral diet (LF-EN) and identical with the half of fat provided by fish oil (FO-EN). Study endpoints: mechanical ventilation time, inflammation (CRP), infectious and other complications, mortality until discharge.

The study is planed as 2 parts: 1) preliminary study testing the feasibility of the study, 2) the study completed with information from the preliminary phase, both phases being randomised and controlled.

DETAILED DESCRIPTION:
Randomisation within the first 24 hours of admission to 2 types of enteral feeds: 1) ω 3 PUFA (FO-EN) or 2) control solution which is the hospitals standard low 18% fat containing solution.

The patients are fed as long as clinically required with the initial solution.

ELIGIBILITY:
Inclusion Criteria:

- adult >16 years, burns > 15% BSA, mechanical ventilation, next of kin consent

Exclusion Criteria:

* absence of the above, absence of commitment to full treatment
* comorbidities (cancer, COPD, diabetes, liver failure (Child Pugh B and C)
* pregnancy

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Number of infections | up to Day 28 after burn injury
  Infectious complications will be recorded according to CDC criteria, and grouped as pulmonary, blood stream infections (catheter related or not), cutaneous, abdominal and others

SECONDARY OUTCOMES:
Non infectious complications | up to day 28
  Any complication will be recorded during the above time frame

OTHER OUTCOMES:
Duration of mechanical ventilation | up to day 28
  Time on mechanical ventilation though an endotracheal tube (naso-tracheal or tracheostomy)
Length of ICU and hospital stay | up to day 28
  ICU and hospital to discharge but maximum for 28 days
Mortality | Hospital stay
Magnitude of CRP increase | during ICU stay and up to day 28
  C-reactive protein as determined for clinical purpose, Temperature (maximal T° per day), Leucocytes

CONTACTS AND LOCATIONS:
Overall Officials: Serrana Tihista, RD, Principal Investigator — Universidad de la República Oriental del Uruguay
Locations (1):
- Centro National de Quemados, Montevideo, Uruguay

REFERENCES:
- [Derived] Tihista S, Echavarria E. Effect of omega 3 polyunsaturated fatty acids derived from fish oil in major burn patients: A prospective randomized controlled pilot trial. Clin Nutr. 2018 Feb;37(1):107-112. doi: 10.1016/j.clnu.2017.01.002. Epub 2017 Jan 16. PMID 28153504